CLINICAL TRIAL: NCT05419193
Title: Efficacy and Safety of Propranolol for the Post-Stroke Pneumonia
Brief Title: PROpranolol for Cerebral Hemorrhage-ASsociated pnEumonia (PRO-CHASE)
Acronym: PRO-CHASE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2022-05-07-001
Record Dates: First submitted 2022-06-02; First posted 2022-06-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Vascular Accident; Intracranial Hemorrhages; Intracerebral Hemorrhage; Hemorrhagic Stroke; Stroke, Acute
Keywords: Stroke; propranolol; infection; treatment
MeSH Terms: conditions — Stroke; Intracranial Hemorrhages; Cerebral Hemorrhage; Hemorrhagic Stroke; Infections | interventions — Propranolol; Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Patients will receive usual care and drug use in hospital.
  Interventions: Other: control group
- Propranolol group (Experimental): Propranolol hydrochloride will be administered intravenously via pump at a initial dose of 5mg/day over a course of 7 consecutive days after randomization.
  Interventions: Drug: Propranolol Hydrochloride

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Day of randomization:
  propranolol IV vp for 7 days after randomization
  Arms: Propranolol group
Other: control group — Patients will receive usual care and drug use in hospital
  Arms: Control group

SUMMARY:
Stroke-associated pneumonia (SAP) is a grave complication of stroke and one of the most important predictors for patients' poor outcomes. Stroke associated pneumoniaSAP and other infections limited the overall efficacy of stroke management. Increasing evidence suggests that sympathetic nervous system activity contributes to post post-stroke immunosuppression and emergence of infections. This study is designed to test the safety and efficacy of an adrenergic β receptor blocker propranolol in reducing SAP in hemorrhagic stroke patients, in a multi-center, randomized, open-labeled, end point-blinded, trial.

DETAILED DESCRIPTION:
This study will enroll 168 intracerebral hemorrhage patients who meet the inclusion criteria.

ICH patients meet the inclusion criteria will be randomly assigned at a 1:1 ratio into groups of standard treatment (blank-controlled), or propranolol hydrochloride injection .

Patients allocated to experimented group will be intravenously given initial dose at 5mg propranolol hydrochloride daily over a course of 7 consecutive days, The primary purpose of this study is to compare propranolol hydrochloride with standard treatment on reducing the 7-day risk of pneumonia when initiated within 24 hours of symptom onset in intracerebral hemorrhage.

Both intent analysis (ITT) and per-protocol (PP) were used for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years older and less than 80 years.
2. Onset of new neurological deficits within≤24 hours at the time of randomization
3. CT scan demonstrates supratentorial parenchymal hemorrhage and volume of hematoma≥10ml .
4. Initial NIHSS score of 11 or greater and less than 25 scores.
5. Initial GCS score (aggregate of verbal, eye, and motor response scores) of 8 or greater at time of enrollment.
6. Admission without infection signs.
7. Signed and dated informed consent by the subject, legally authorized representative, or surrogate obtained.

Exclusion Criteria:

1. Subjects is considered a candidate for immediate surgical intervention by the neurosurgery service, including surgical evacuation of hematoma, decompressive craniectomy, minimally invasive aspiration of hematoma, and ventricular shunt or external ventricular drainage for intracerebral hemorrhage into the ventricle.
2. Patients with primary intraventricular hemorrhage or cerebral hemorrhage due to a definite cause, such as trauma, vascular malformation, aneurysm, coagulopathy, anticoagulant or antiplatelet drugs, thrombolytic therapy, post-infarction hemorrhagic transformation, hematologic disease, moyamoya disease, primary or metastatic tumor, venous sinus thrombosis, vasculitis, etc.
3. Previous stroke or pre-onset motor disability (mRS≥1)
4. Pregnancy or parturition within previous 30 days or active lactation.
5. Use of beta blockers (propranolol, metoprolol, sotalol, carvedilol, bisoprolol, atenolol, esmolol, etc.) or reserpine within the last 30 days.
6. Bronchial asthma or chronic obstructive pulmonary disease
7. Cardiogenic shock or severe or acute heart failure.
8. Degree II-III atrioventricular block or sinus bradycardia or heart rate ≤65/min.
9. Known sensitivity to propranolol.
10. Severe hepatic or renal insufficiency
11. History of Malignancy
12. Currently participating in other interventional clinical trials.
13. Immunosuppressant therapy or known immunosuppression.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Incidence of stroke-associated pneumonia | up to 7days
  Stroke-associated pneumonia diagnosed in accordance to a defined algorithm.

SECONDARY OUTCOMES:
Clinical improvement | up to 90 days
  Modified Rankin Scale （mRS，0-6 scores, poor outcome defined as mRS≥4）are used to describe the clinical improvement at baseline, 7days, 14days, 30days and 90days.
Change in immunology function [ Time Frame: up to 7 days ]（ONLY patients recruited from Beijing Tiantan hospital and Tangdu Hospital, Air Force Medical University will receive this evaluation） | up to 7 days
  Use the flow cytometry to measure the change of ratio and number of CD4+、CD8+、NK 、B cells at baseline, 3 days, 7 days
Spleen volume [ Time Frame: up to 7 days ] （ONLY patients recruited from Beijing Tiantan hospital and Tangdu Hospital, Air Force Medical University will receive this evaluation） | up to 7 days
  Spleen volume calculated based on Abdominal CT.
Adverse Event (AE) | up to 90 days
  Per protocol Adverse Event (AE), Adverse Reaction (AR), Serious Adverse Event / Reaction (SAE / SAR), and Suspected Unexpected Serious Adverse Reactions (SUSAR)

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Lu'an Hospital of Traditional Chinese Medicine, Lu'an, Anhui
  - Beijing Tiantan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Third Affiliated Hospital, Soochow University, Changzhou, Jiangsu
  - Weinan City Center hospital, Weinan, Shaanxi
  - Tangdu Hospital,Air Force Medical University, Xi'an, Shaanxi
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Qianxian People's Hospital, Xianyang, Shaanxi
  - The First People' Hospital of Xian Yang, Xianyang, Shaanxi
  - Xianyang hospital affliated of Yan'an University, Xianyang, Shaanxi
  - The 970th Hospital of the Chinese People's Liberation Army (Weihai Branch), Weihai, Shandong
  - The 970th Hospital of the Chinese People's Liberation Army (Yantai Branch), Yantai, Shandong
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
The study protocol,statistical analysis plan(SAP),informed consent form(ICF),clinical study report(CSR),analytic code will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code